CLINICAL TRIAL: NCT01970722
Title: Cytoreductive Surgery With Hyperthermic Intraperitoneal Chemotherapy (HIPEC) and Optional Postoperative Normothermic Intraperitoneal (IP) Chemotherapy to Treat Primary or Recurrent Carcinoma of Ovarian, Fallopian Tube, Uterine, or Peritoneal Origin
Brief Title: Surgery and Chemotherapy With or Without Chemotherapy After Surgery in Treating Patients With Ovarian, Fallopian Tube, Uterine, or Peritoneal Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12316; NCI-2013-01948 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 122550; 108303; 116613; 122035; 12316 (Other: City of Hope Medical Center)
Record Dates: First submitted 2013-10-23; First posted 2013-10-28 (Estimated); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: FIGO Stage IVA Ovarian Cancer; FIGO Stage IVB Ovarian Cancer; Platinum-Resistant Ovarian Carcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma; Recurrent Uterine Corpus Carcinoma; Stage III Fallopian Tube Cancer AJCC v7; Stage III Ovarian Cancer AJCC v6 and v7; Stage III Primary Peritoneal Cancer AJCC v7; Stage III Uterine Corpus Cancer AJCC v7; Stage IIIA Fallopian Tube Cancer AJCC v7; Stage IIIA Ovarian Cancer AJCC v6 and v7; Stage IIIA Primary Peritoneal Cancer AJCC v7; Stage IIIA Uterine Corpus Cancer AJCC v7; Stage IIIB Fallopian Tube Cancer AJCC v7; Stage IIIB Ovarian Cancer AJCC v6 and v7; Stage IIIB Primary Peritoneal Cancer AJCC v7; Stage IIIB Uterine Corpus Cancer AJCC v7; Stage IIIC Fallopian Tube Cancer AJCC v7; Stage IIIC Ovarian Cancer AJCC v6 and v7; Stage IIIC Primary Peritoneal Cancer AJCC v7; Stage IIIC Uterine Corpus Cancer AJCC v7; Stage IV Fallopian Tube Cancer AJCC v6 and v7; Stage IV Ovarian Cancer AJCC v6 and v7; Stage IV Primary Peritoneal Cancer AJCC v7; Stage IV Uterine Corpus Cancer AJCC v7; Stage IVA Uterine Corpus Cancer AJCC v7; Stage IVB Uterine Corpus Cancer AJCC v7
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Gemcitabine; Paclitaxel; Taxes; liposomal doxorubicin; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (surgery, HIPEC cisplatin) (Experimental): Patients undergo surgery and receive hyperthermic cisplatin IP over 60 minutes.
  Beginning at least 3 weeks after surgery, patients may receive carboplatin, paclitaxel, pegylated liposomal doxorubicin hydrochloride, or gemcitabine hydrochloride IP or IV at the discretion of the medical and gynecologic oncologists.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Gemcitabine Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Drug: Pegylated Liposomal Doxorubicin Hydrochloride; Other: Quality-of-Life Assessment; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Carboplatin — Given IP or IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cisplatin — Given IP
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone''s Chloride; Peyrone''s Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Gemcitabine Hydrochloride — Given IP or IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; FF 10832; FF-10832; FF10832; Gemcitabine HCI; Gemzar; LY-188011; LY188011
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IP or IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Drug: Pegylated Liposomal Doxorubicin Hydrochloride — Given IP or IV
  Other Names: ATI-0918; Caelyx; DOX-SL; Doxil; Doxilen; Doxorubicin HCl Liposomal; Doxorubicin HCl Liposome; Doxorubicin Hydrochloride Liposome; Duomeisu; Evacet; LipoDox; Lipodox 50; Liposomal Adriamycin; liposomal doxorubicin hydrochloride; Liposomal-Encapsulated Doxorubicin; Pegylated Doxorubicin HCl Liposome; S-Liposomal Doxorubicin; Stealth Liposomal Doxorubicin; TLC D-99
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Procedure: Therapeutic Conventional Surgery — Undergo surgery

SUMMARY:
This phase I trial studies the side effects and how well surgery and heated chemotherapy with or without non-heated chemotherapy after surgery works in treating patients with ovarian, fallopian tube, uterine, or peritoneal cancer. Giving a dose of heated chemotherapy into the abdomen during surgery that is done to remove ovarian, fallopian tube, uterine, or peritoneal cancer may help lower the risk of the cancer coming back. Giving unheated chemotherapy drugs directly into the abdomen after surgery may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether cytoreductive surgery with hyperthermic intraperitoneal chemotherapy (HIPEC) followed by postoperative normothermic intraperitoneal (IP) chemotherapy is feasible and safe to administer, as measured by toxicities occurring during treatment or follow-up.

SECONDARY OBJECTIVES:

I. To determine quality of life (QoL) and compare the outcomes to a historical control of IP chemotherapy (no HIPEC) for women with ovarian cancer.

II. To determine whether cytoreductive surgery with HIPEC alone is feasible and safe to administer, as measured by toxicities occurring during treatment or follow-up.

III. To estimate progression-free survival (PFS). IV. To collect biospecimens and perform correlative translational studies focused on understanding the mechanisms of action of HIPEC on ovarian cancer.

OUTLINE:

Patients undergo surgery and receive hyperthermic cisplatin intraperitoneally (IP) over 60 minutes.

Beginning at least 3 weeks after surgery, patients may receive carboplatin, paclitaxel, pegylated liposomal doxorubicin hydrochloride, or gemcitabine hydrochloride IP or intravenously (IV) at the discretion of the medical and gynecologic oncologists.

After completion of study treatment, patients are followed up at 3-6, 6-9, 9-12, and 12-15 months; every 3 months for 1 year; and then every 4 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Provided informed consent
* Patient with primary or recurrent International Federation of Gynecology and Obstetrics (FIGO) stage III or IV, or recurrent ovarian, fallopian tube, peritoneal carcinoma, or uterine cancer, confined to abdominal cavity, including those who have completed neoadjuvant chemotherapy and primary surgery
* Gynecologic Oncology Group (GOG) or Eastern Cooperative Oncology Group (ECOG) performance status =< 1 or Karnofsky scale (KPS) >= 70%
* Patients who are platinum-sensitive or platinum resistant
* Candidate for potentially radical, maximal effort cytoreductive surgery at the discretion and expertise of the treating physician
* For patients with newly diagnosed-ovarian/tubal/peritoneal cancer who have received pre-operative neoadjuvant chemotherapy, evidence of response must be documented by at least one of the following:

  * Decline in serum cancer antigen (CA) 125 level
  * At least a 30% decrease in the sum of the longest diameter of target lesions on radiographic imaging
  * Improvement of ascites volume
  * Neoadjuvant chemotherapy must be held for at least 3 weeks prior to surgery
  * Resolution of any effects of prior therapy (except alopecia and peripheral neuropathy) to the current National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (NCI CTCAE) grade =< 1 and to baseline laboratory values as defined
* Hemoglobin (HGB) >= 9 g/dL
* White blood cell (WBC) >= 3,000/mcL
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets (PLT) >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Serum glutamic oxaloacetic transaminase (SGOT)/serum glutamate pyruvate transaminase (SGPT) < 2.5 x institutional upper limit of normal (ULN)
* Creatinine < 1.5 x ULN or creatinine clearance > 60 ml/min according to Cockcroft-Gault formula
* Neuropathy (sensory and motor) NCI CTCAE grade =< 2
* Prothrombin time (PT) such that international normalized ratio (INR) is < 1.5 (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin or low molecular weight heparin) and a partial thromboplastin time (PTT) < 1.2 times control
* Serum albumin >= 2.5
* No active infection requiring antibiotics
* Preoperative or intraoperative (frozen section) diagnosis of ovarian, peritoneal, fallopian tubal or uterine cancer
* Surgery achieves either no gross residual disease (R0) or optimal cytoreductive status defined as no single lesion measuring more than 5.0 mm in its greatest diameter
* Stable from a cardiopulmonary standpoint to continue with prolonged surgery and anesthesia

Exclusion Criteria:

* Patients with active extra-abdominal disease including active malignant pleural effusion; patients who have been successfully treated with neoadjuvant chemotherapy and no longer have (malignant) pleural effusions may be included
* Patients whose disease has progressed following at least 3 cycles of neoadjuvant chemotherapy as defined by at least one of the following:

  * Doubling of serum CA-125 level
  * At least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions
  * Clinical deterioration (worsening ascites, carcinomatous ileus, malignant bowel obstruction, severe hypoalbuminemia, declining performance status)
* Cardiac or pulmonary conditions that preclude aggressive cytoreductive surgery
* Patients whose circumstances do not permit completion of the study or the required follow-up
* Pregnant, nursing, or of childbearing potential and refuse hysterectomy or bilateral salpingo-oophorectomy
* Other active invasive malignancies, with the exception of non-melanoma skin cancer and breast cancer (if without evidence of disease 1 year after completion of treatment)
* Metastatic non-gynecologic or breast primaries
* Sub-optimal resection as their surgical outcome
* Intraoperative frozen section suggesting hepatobiliary, pancreatic, adrenal, or urinary tract cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-05-19 (Actual); Primary Completion 2026-02-03 (Estimated); Study Completion 2026-02-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related toxicities according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) guidelines | Up to 3 months post-surgery
  Toxicity for both primary and recurrent groups will be summarized using frequency tables.

SECONDARY OUTCOMES:
Quality of life (QoL) assessed by the Functional Assessment of Cancer Therapy-Ovarian (FACT-O) QoL questionnaire | Up to 15 months post-surgery
  The FACT-O has four subscales: physical, social/family, emotional, and functional well-being. Answers are on a scale of 0 'not at all' to 4 'very much'. To estimate effect sizes over time, generalized linear models will be used to estimate the correlations between potential prognostic factors. Generalized estimating equations (GEEs) have utility in modeling longitudinal effects across time in prospective cohorts, and the models will include time-dependent covariate structures for continuous outcomes. QoL will be compared to a historical control of intraperitoneal (IP) chemotherapy for women with ovarian cancer.
Progression-free survival (PFS) | From time-of-study entry to time-of-detection of new lesions on computed tomography imaging that is triggered by CA125 progression as defined by Gynecologic Cancer Intergroup Criteria (GCIG) or clinical symptoms or deterioration, assessed up to 3 years
  PFS will be estimated in both groups. The survival curve will be estimated using Kaplan-Meier method and graphically displayed along with the corresponding 95% confidence curves. The Cox proportional hazards model will be used to derive an estimate of the hazard ratio and its corresponding 95% confidence limits.

CONTACTS AND LOCATIONS:
Overall Officials: Thanh Dellinger, Principal Investigator — City of Hope Medical Center
Locations (4):
- United States (4):
  - City of Hope Corona, Corona, California
  - City of Hope Medical Center, Duarte, California
  - City of Hope Upland, Upland, California
  - Parkview Hospital Randallia, Fort Wayne, Indiana

REFERENCES:
- [Derived] Dellinger TH, Han ES, Raoof M, Lee B, Wu X, Cho H, He TF, Lee P, Razavi M, Liang WS, Schmolze D, Priceman SJ, Lee S, Lin WC, Lin JF, Kebria M, Hakim A, Ruel N, Stewart DB, Wang EW, Paz BI, Wakabayashi MT, Cristea MC, Rodriguez-Rodriguez L. Hyperthermic Intraperitoneal Chemotherapy-Induced Molecular Changes in Humans Validate Preclinical Data in Ovarian Cancer. JCO Precis Oncol. 2022 Mar;6:e2100239. doi: 10.1200/PO.21.00239. PMID 35357903